CLINICAL TRIAL: NCT06695676
Title: Evaluation of Left Ventricle Systolic Functions of Patients On Lurasidone
Brief Title: Effects of Lurasidone on Left Ventricle Systolic Functions
Acronym: Lurasidone
Status: Not yet recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sevil Gulastı, Cardiologist, Aydin Adnan Menderes University
Other Study IDs: 2024/164
Record Dates: First submitted 2024-11-17; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Lurasidone Cardiotoxicity; Schizophrenia Patients; Bipolar Disorders
Keywords: Global Longitudinal Strain; Cardiotoxicity; Lurasidone; antipsychotic drugs
MeSH Terms: conditions — Bipolar Disorder; Cardiotoxicity | interventions — Global Longitudinal Strain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients on Lurasidone: Patient who are admitted by the psychiatry clinic of our center and meet the inclusion criteria
  Interventions: Diagnostic Test: Global Longitudinal Strain

INTERVENTIONS:
Diagnostic Test: Global Longitudinal Strain — Global longitudinal strain measurement is a more objective method to determine left ventricular systolic function than traditional eyeballing method. It helps to detect and quantify subtle changes even so it is an emerging method to evaluate the cardiotoxicity of chemotherapeutic drugs. It is planned to compare each selected patient's GLS measurement before starting to use lurasidone and after six months of using it. Hereby our aim is to find if lurasidone has any effect on left ventricular systolic function.

SUMMARY:
The goal of our study to learn if lurasidone molecule which is used on patients with schizophrenia or bipolar disorder has any cardiotoxic effect.

DETAILED DESCRIPTION:
Lurasidone is an atypical antipsychotic drug used both on patients with schizophrenia or bipolar disorder. It improves patients' clinical symptoms through dopamine D2 and serotonin 5-HT2A receptor antagonism. However, the effect of antipsychotic drugs on cardiac functions is an important parameter for patient safety during the treatment process. Although the existing literature on the cardiac effects of lurasidone is limited, atypical antipsychotic are known to cause corrected QT interval prolongation, arrhythmias and suppression on cardiac functions. Studies show that these cardiac side effects are mostly related to clozapine which is a D2 and 5-HT2A antagonist such as lurasidone. Though not fully understood, it is thought that cardiac events due to antipsychotic drugs occur because of type 1 hypersensitivity and rising levels of pro-inflammatory cytokines. It might also be related to ischemia that free oxygen radicals initiate at the molecular level.

D2 receptors play a critical role in the regulation of heart rate and vascular tone. D2 receptor antagonism may increase the risk of hypertension by changing systemic vascular resistance and heart rate. In addition, inhibition of D2 receptors may lead to loss of the vasodilator effects of dopamine, leading to impaired cardiovascular homeostasis. Similarly 5-HT2A receptors have important effects of cardiac functions. 5-HT2A receptor antagonism, together with imbalances in serotonin levels, may increase heart rate and affect vascular tone, leading to vasoconstriction. It is possible that the increase in systemic vascular resistance and cardiac inotropy through receptor antagonism may cause deterioration in cardiac functions and should be considered in clinical follow-up.

There are a limited number of studies examining the potential effects of lurasidone on cardiac functions. For example, one study reported that lurasidone treatment did not cause a significant prolongation of the QTc interval, while another study reported that the overall cardiac safety profile of lurasidone use was quite favorable. However, more data are needed to compare cardiac side effects between lurasidone and other antipsychotics and how these effects should be managed in clinical practice. The aim of this study is to gain information about the possible cardiac effects of the lurasidone molecule by evaluating left ventricular systolic function with the help of periodic transthoracic echocardiography. In particular, clarifying the potential risks of lurasidone on cardiac health and the clinical significance of these risks is important both to increase patient safety and to optimize treatment processes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Diagnosed with schizophrenia or bipolar disorder by the psychiatry clinic of our center and indicated to use lurasidone molecule
* Hasn't been diagnosed with coronary artery disease, any kind of heart failure or severe valvular disease

Exclusion Criteria:

* Patients who do not agree to participate to the trial
* Patient who do not meet the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who apply to Adnan Menderes University Psychiatry Clinic and meet the criteria of inclusion
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Lurasidone molecule will affect left ventricular systolic function | All patients whom are admitted by our psychiatry clinic for the next 6 months will be included.
  We will measure left ventricular global longitudinal strain of each selected patient before starting to use lurasidone and perform the same evaluation for every patient six months later. Since global longitudinal strain measurement is a preferred way to detect subtle changes of wall motions and contractile functions, we will be able detect if this molecule has any negative effect on left ventricular systolic function.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University, Aydin, Zafer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slawinski G, Hawryszko M, Lizewska-Springer A, Nabialek-Trojanowska I, Lewicka E. Global Longitudinal Strain in Cardio-Oncology: A Review. Cancers (Basel). 2023 Feb 3;15(3):986. doi: 10.3390/cancers15030986. PMID 36765941
- [Background] Alawami M, Wasywich C, Cicovic A, Kenedi C. A systematic review of clozapine induced cardiomyopathy. Int J Cardiol. 2014 Sep 20;176(2):315-20. doi: 10.1016/j.ijcard.2014.07.103. Epub 2014 Aug 1. PMID 25131906
- [Background] Curto M, Girardi N, Lionetto L, Ciavarella GM, Ferracuti S, Baldessarini RJ. Systematic Review of Clozapine Cardiotoxicity. Curr Psychiatry Rep. 2016 Jul;18(7):68. doi: 10.1007/s11920-016-0704-3. PMID 27222142
- See also: How and Why to Use Global Longitudinal Strain Measurement — https://heart.bmj.com/content/106/18/1438